CLINICAL TRIAL: NCT05331560
Title: Efficacy and Safety of Transcranial Pulse Stimulation (TPS) in Older Adults With Mild Neurocognitive Disorder - an Open-label Self-controlled Trial
Brief Title: Transcranial Pulse Stimulation Open-label Self-controlled Trial For Mild Neurocognitive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Storz Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW20-024
Record Dates: First submitted 2022-03-23; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Mild Neurocognitive Disorder
Keywords: Transcranial pulse stimulation; mild neurocognitive disorder; open-label; self-controlled trial
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Masking Description: Since TPS is a new NIBS technology, no studies have been done on older adults with mild NCD, which is a golden period for intervention before the pathology involved the whole brain and leading to irreversible damage. We would like to perform an open-label self-controlled study to assess the effectiveness and tolerability of TPS with neuro-navigation on cognition in older adults with mild NCD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): A 2-week intervention TPS intervention will result in a significant improvement in the Montreal Cognitive Assessment (HK-MoCA; Hong Kong Chinese version), which will be maintained for 12 weeks.
  Interventions: Device: Transcranial Pulse Stimulation (TPS)

INTERVENTIONS:
Device: Transcranial Pulse Stimulation (TPS) — A global brain stimulation approach, which homogenously distributes the total energy of 6000 TPS pulses per session over all accessible brain areas.
  Prefrontal, Temporal and Occipital brain areas were stimulated by ultrashort (3μs) ultrasound pulses with typical energy levels of 0.2-0.25 mJ/mm2 and pulse frequencies of 4-5 Hz (pulses per second).

SUMMARY:
Background:

A significant proportion of older adults suffered from age-related diseases particularly dementia, also known as major neurocognitive disorder (NCD), which is becoming a worldwide health burden. In principle, Interventions for dementia should have optimal benefits at the earliest preclinical stage yet no evidence has been found to support a particular pharmacological approach in preventing cognitive decline during the stage of mild NCD. Non-invasive brain stimulation (NIBS), on the other hand, is increasingly recognized as a potential alternative to tackle this problem. Typical NIBS include transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS). A new kind of NIBS named Transcranial Pulse stimulation (TPS) is also recently used for treating patients with Alzheimer's disease (AD).TPS is a kind of NIBS that uses repetitive sin ultrashort pulses in the ultrasound frequency range to stimulate the brain, and it can provide better spatial precision and reach deeper brain regions comparing to tDCS and TMS. The mechanism of TPS is to convert the mechanical TPS stimulus into biochemical responses, thus influence some fundamental cell functions. A recent study showed that there is a significant improvement in using TPS in treating AD. However, there has been no study investigating the effect of TPS on older adults with mild NCD.

Objective:

This study is an open-label self-controlled study to assess the effectiveness and tolerability of TPS on cognition in older adults with mild NCD. We hypothesized that a 2-week TPS intervention could significantly improve patient's global cognition which will be maintained for 12 weeks.

Design:

The current study is an open-label self-controlled interventional trial of TPS guided by neuro-navigation using structural MRI. All participants will undergo the treatment as usual (TAU) period as self-controlled for 12 weeks. They will then receive a six-session TPS intervention for 2 weeks with three sessions per week. A 12 weeks post-intervention assessment will then be conducted.

Data Analysis:

Primary outcome and secondary outcomes assessment would be carried out at baseline, after TAU period, immediately after the intervention and 12 weeks after the intervention. The primary outcome will be the change of the Hong Kong Chinese version of the Montreal Cognitive Assessment (HK-MoCA). The secondary outcome includes specific cognitive domains, daily functioning, mood, and apathy. The intention-to-treat analysis would be carried out.

Significance:

The result of the current study would provide further data on the effectiveness and tolerability of TPS as a new treatment in patients with mild NCD.

DETAILED DESCRIPTION:
Background Age-related diseases, particularly dementia, now known as major neurocognitive disorder (NCD), are a great health burden in Hong Kong and worldwide. Interventions that aim to ameliorate cognitive decline or prevent dementia offer a compelling alternative paradigm for reducing the impact of the disease, not only on individuals but also on their families and on society. In principle, to achieve its optimal benefits, intervention for dementia should begin at the earliest preclinical stage. However, no evidence has been found to support a pharmacological approach to the prevention, reduction, or postponement of cognitive decline during the stage of mild NCD. Besides pharmacological approaches, non-invasive brain stimulation (NIBS) is increasingly recognised as a potential alternative to tackle this problem. The typical examples of NIBS are transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS). Besides these, there is a new NIBS named transcranial pulse stimulation (TPS), also known as low-intensity extracorporeal shock wave therapy (Li-ESWT), which recently obtained CE marking in 2018 for the treatment of the central nervous system (CNS) in patients with mild to moderate Alzheimer's disease (AD).

The introduction of TPS TPS is using repetitive single ultrashort pulses in the ultrasound frequency range to stimulate the brain. With a neuro-navigation device, TPS can achieve this in a highly focal and precisely targeted manner. TPS differs from tDCS and TMS using direct or induced electric current. Using electric current to stimulate the brain may be limited by the problem of conductivity and failure to reach deep brain regions. Instead, low-intensity focused ultrasound provides good spatial precision and resolution to noninvasively modulate subcortical areas, despite the problem of skull attenuation. Using lower ultrasound frequencies TPS can successfully improve skull penetration in humans.

Biological mechanism of TPS The basic mechanism of TPS is mechanotransduction. It is a biological pathway through which the cells convert the mechanical TPS stimulus into biochemical responses, thus influencing some fundamental cell functions such as migration, proliferation, differentiation, and apoptosis. The ultrashort ultrasound pulse could enhance the cell proliferation and differentiation in cultured neural stem cell, which plays an important role in the repair of brain function in CNS diseases. The TPS may affect neurons and induce neuroplastic effects through several pathways including increasing cell permeability, stimulation of mechanosensitive ion channels, the release of nitric oxide resulting in vasodilation, increased metabolic activity and angiogenesis, stimulation of vascular growth factors (VEGF) and stimulation of brain derived neurotrophic factor (BDNF).

Clinical effects of TPS Focused ultrasound demonstrated the neuromodulation effect in the human brain. Focused ultrasound can modulate the amplitude of somatosensory evoked potentials (SEPs) when targeted at the cortical regions that generate these potentials and even the deep structure such as the thalamus. TPS, previously named as Li-ESWT was applied to five patients with unresponsive wakefulness syndrome. They received 4-week (3 times per week) treatment, 4000 pulses each, every 6 months for an average of two to four years. There was significant improvement in the vigilance and in three patients the percutaneous endoscopic gastrostomy (PEG) tube could be removed due to improved oropharyngeal motor function. In the most recent study, TPS was applied to 35 elderly with AD. They were treated in 3 TPS sessions (6000 pulses each) per week for 2-4 weeks, either over classical AD affected sites such as the dorsolateral prefrontal cortex, areas of the memory and language network, or over all accessible brain areas (global brain stimulation). Significant improvement in the CERAD (Consortium to Establish a Registry for Alzheimer's Disease) score was demonstrated (immediately as well as 1 and 3 months after stimulation. fMRI also showed significant increased connectivity within the memory network.

Safety issue of TPS TPS uses very low energy for the brain stimulation. In vivo animal TPS study did not cause any tissue damage despite using 6-7-fold higher energy levels compared with those in human studies. Furthermore, the intervention did not cause any serious adverse effects such as intracranial bleeding, oedema or other intracranial pathology, as confirmed with MRI in a previous AD study. Few subjects reported headache (4%), pain or pressure (1%) and mood deterioration (3%). The CE marked TPS system has proven to be safe in >1500 treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1. 60 years of age or above
* 2. Chinese ethnicity
* 3. Mild neurocognitive disorder (NCD) meeting the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria
* 4. At least 3 months of stable anti-dementia therapy prior to enrolment (unchanged medication, if receiving)
* 5. Written informed consent

Exclusion Criteria:

* 1. A HK-MoCA score below the second percentile according to the subject's age and education level
* 2. Alcohol or substance dependence
* 3. Concomitant unstable major medical conditions or major neurological conditions such as brain tumour, brain aneurysm
* 4. Haemophilia or other blood clotting disorders or thrombosis
* 5. Significant communicative impairments
* 6. Participants with any metal implant in brain or treated area of the head

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Global Cognition | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Global cognition measured using the Hong Kong Chinese version of the Montreal Cognitive Assessment (HK-MoCA) is our primary outcome. The total score ranges from 0-30 with higher scores indicating better cognition.

SECONDARY OUTCOMES:
Changes in Verbal Fluency | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Measured by the category verbal fluency test.
Change in Working Memory | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Measured by forward and backward digit span test.
Change in Executive Functioning | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Measured by the Trail Making Test Parts A and B.
Change in Attention | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Measured by the Stroop test.
Change in Depressive Symptoms | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Depressive symptoms will be assessed by the HAM-D-17, which is a widely used and reliable measure of depressive symptoms. Scores range from 0 to 52, with higher scores indicating more severe depression.
Change in Daily Functioning | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  Instrumental activities of daily living will be assessed with the Hong Kong Chinese version of the Lawton Instrumental Activities of Daily Living Scale.
Change in Apathy | Baseline, 12-week Treatment-As-Usual, Immediate after 2-week TPS Treatment, 12-week Follow-up
  The severity of apathy will be measured using the Hong Kong version of the Apathy Evaluation Scale (AES-HK) (in press, abstract). The AES-HK is an 18-item scale designed to measure apathy as a neuropsychiatric symptom. It is the most psychometrically sound measure of apathy across some disease populations. The internal consistency of the AES-HK was estimated using Cronbach's alpha, which yielded a coefficient of 0.946. The inter-rater and test-retest reliability were both satisfactory.
Change in Adverse Effects and Risk Indicators | Across 6 TPS Treatment sessions
  A checklist of potential adverse effects associated with TPS administration will be generated from the available literature on AD. The checklist will be used to monitor tolerability and adverse events in each session throughout the intervention.
Changes in Brain Regional Volume Differences and White Matter Hyperintensities (WMH) | Baseline, 12-week Follow-up
  Participants will receive pre and post treatment MRI scan to measure any changes in structural and functional connectivity changes in the brain. Structural MRI scans including T1- and T2-weighted fluid attenuation inversion recovery (T2-FLAIR) sequences, and Diffusion tensor imaging (DTI) will be used for assessing regional volume differences and WMH across the whole brain.
Change in Brain Functional Connectivity | Baseline, 12-week Follow-up
  Participants will receive pre and post treatment MRI scan to measure any changes in structural and functional connectivity changes in the brain. Resting-state fMRI of 150 T2-weighted gradient echo planar imaging (EPI) will be acquired, during which subjects will view a fixation cross ('+') passively at the centre of the screen. All resting state-fMRI (rs-fMRI) volumes will be pre-processed, with motion correction, slice timing correction, then linearly registered to the Montreal Neurological Institute (MNI) standard space.
Change in Brain-Derived Neurotrophic Factor (BDNF) | Baseline, Immediate after 2-week TPS Treatment
  A 20 ml venous blood sample will be collected from all participants before and after the TPS intervention to examine Brain-derived neurotrophic factor (BDNF).

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Pak Wing Cheng, MBBS (HKU), Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Jockey Club Building for Interdisciplinary Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Since the study involves sensitive and private medical history from recruited or self-enrolled subjects, individual data will not be available to other researchers.

REFERENCES:
- [Background] Beisteiner R, Matt E, Fan C, Baldysiak H, Schonfeld M, Philippi Novak T, Amini A, Aslan T, Reinecke R, Lehrner J, Weber A, Reime U, Goldenstedt C, Marlinghaus E, Hallett M, Lohse-Busch H. Transcranial Pulse Stimulation with Ultrasound in Alzheimer's Disease-A New Navigated Focal Brain Therapy. Adv Sci (Weinh). 2019 Dec 23;7(3):1902583. doi: 10.1002/advs.201902583. eCollection 2020 Feb. PMID 32042569
- [Background] d'Agostino MC, Craig K, Tibalt E, Respizzi S. Shock wave as biological therapeutic tool: From mechanical stimulation to recovery and healing, through mechanotransduction. Int J Surg. 2015 Dec;24(Pt B):147-53. doi: 10.1016/j.ijsu.2015.11.030. Epub 2015 Nov 28. PMID 26612525
- [Background] Hatanaka K, Ito K, Shindo T, Kagaya Y, Ogata T, Eguchi K, Kurosawa R, Shimokawa H. Molecular mechanisms of the angiogenic effects of low-energy shock wave therapy: roles of mechanotransduction. Am J Physiol Cell Physiol. 2016 Sep 1;311(3):C378-85. doi: 10.1152/ajpcell.00152.2016. Epub 2016 Jul 13. PMID 27413171
- [Background] Ingber DE. Cellular mechanotransduction: putting all the pieces together again. FASEB J. 2006 May;20(7):811-27. doi: 10.1096/fj.05-5424rev. PMID 16675838
- [Background] Legon W, Ai L, Bansal P, Mueller JK. Neuromodulation with single-element transcranial focused ultrasound in human thalamus. Hum Brain Mapp. 2018 May;39(5):1995-2006. doi: 10.1002/hbm.23981. Epub 2018 Jan 29. PMID 29380485
- [Background] Legon W, Sato TF, Opitz A, Mueller J, Barbour A, Williams A, Tyler WJ. Transcranial focused ultrasound modulates the activity of primary somatosensory cortex in humans. Nat Neurosci. 2014 Feb;17(2):322-9. doi: 10.1038/nn.3620. Epub 2014 Jan 12. PMID 24413698
- [Background] Lohse-Busch H, Reime U, Falland R. Symptomatic treatment of unresponsive wakefulness syndrome with transcranially focused extracorporeal shock waves. NeuroRehabilitation. 2014 Jan 1;35(2):235-44. doi: 10.3233/NRE-141115. PMID 24990026
- [Background] Mariotto S, Cavalieri E, Amelio E, Ciampa AR, de Prati AC, Marlinghaus E, Russo S, Suzuki H. Extracorporeal shock waves: from lithotripsy to anti-inflammatory action by NO production. Nitric Oxide. 2005 Mar;12(2):89-96. doi: 10.1016/j.niox.2004.12.005. PMID 15740982
- [Background] Minjoli S, Saturnino GB, Blicher JU, Stagg CJ, Siebner HR, Antunes A, Thielscher A. The impact of large structural brain changes in chronic stroke patients on the electric field caused by transcranial brain stimulation. Neuroimage Clin. 2017 Apr 18;15:106-117. doi: 10.1016/j.nicl.2017.04.014. eCollection 2017. PMID 28516033
- [Background] Spagnolo PA, Wang H, Srivanitchapoom P, Schwandt M, Heilig M, Hallett M. Lack of Target Engagement Following Low-Frequency Deep Transcranial Magnetic Stimulation of the Anterior Insula. Neuromodulation. 2019 Dec;22(8):877-883. doi: 10.1111/ner.12875. Epub 2018 Oct 29. PMID 30370983
- [Background] Raschetti R, Albanese E, Vanacore N, Maggini M. Cholinesterase inhibitors in mild cognitive impairment: a systematic review of randomised trials. PLoS Med. 2007 Nov 27;4(11):e338. doi: 10.1371/journal.pmed.0040338. PMID 18044984
- [Background] Wang B, Ning H, Reed-Maldonado AB, Zhou J, Ruan Y, Zhou T, Wang HS, Oh BS, Banie L, Lin G, Lue TF. Low-Intensity Extracorporeal Shock Wave Therapy Enhances Brain-Derived Neurotrophic Factor Expression through PERK/ATF4 Signaling Pathway. Int J Mol Sci. 2017 Feb 16;18(2):433. doi: 10.3390/ijms18020433. PMID 28212323
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] Zhang J, Kang N, Yu X, Ma Y, Pang X. Radial Extracorporeal Shock Wave Therapy Enhances the Proliferation and Differentiation of Neural Stem Cells by Notch, PI3K/AKT, and Wnt/beta-catenin Signaling. Sci Rep. 2017 Nov 10;7(1):15321. doi: 10.1038/s41598-017-15662-5. PMID 29127399